CLINICAL TRIAL: NCT04757571
Title: The GRK2 Inhibitor Paroxetine as a Novel Adjunct to Conventional Therapy in Rheumatoid Arthritis Patients. A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial.
Brief Title: The GRK2 Inhibitor Paroxetine as a Novel Adjunct to Conventional Therapy in Rheumatoid Arthritis Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RS10/2021
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paroxetine (Experimental): Paroxetine 20 mg daily plus standard therapy
  Interventions: Drug: Paroxetine
- Placebo (Placebo Comparator): Placebo tablet daily plus standard therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paroxetine — Paroxetine 20 mg tablet plus standard therapy
  Arms: Paroxetine
Drug: Placebo — Placebo tablet plus standard therapy
  Arms: Placebo

SUMMARY:
Among three MAPK families, paroxetine was found to be able to decrease the phosphorylation of ERK. It was reported that paroxetine attenuates the symptoms of collage induced arthritis rats due to its inhibitory effect on T cell activation and infiltration to synovial tissue via suppression of ERK pathway. This study aimed to evaluate the therapeutic efficacy of paroxetine in rheumatoid arthritis. Paroxetine prevents the joint inflammation which is at the very early stage. paroxetine could inhibit GRK2 with selectivity over other GRKs. Medications developed for maintaining the immunologic equilibrium. such as GRK2 inhibitors, will be the novel trends in RA treatment that could avoid the adverse side effects that are common with current treatment options.

ELIGIBILITY:
Inclusion Criteria:

• Patients with active rheumatoid arthritis based on DAS28 score. Patients received the standard therapy (i.e. one or more conventional DMARDs) for at least three months.

Exclusion Criteria:

* Known hypersensitivity to metformin.
* Patients who have a prior diagnosis with diabetes mellitus.
* Patients receive metformin for any other indications.
* Patients with congestive heart failure.
* Patients with a history of myocardial infarction.
* Patients with severe anemia.
* Patients with active infections or other inflammatory diseases.
* Patients receiving biological therapy.
* Pregnancy or lactation.
* Patients with impaired liver functions.
* Patients with impaired kidney functions (serum creatinine concentrations ≥1.5 and ≥1.4 mg/dL in males and females respectively).
* Patients with malignancies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ACR 20% improvement criteria (ACR20) response rate | week 12
  based on tender and swollen joint counts, patient's assessment of pain, patient and physician global assessment of arthritis, Health Assessment Questionnaire Disability Index (HAQ DI), and CRP level
ACR50 & ACR70 response rate | week 12
  based on tender and swollen joint counts, patient's assessment of pain, patient and physician global assessment of arthritis, Health Assessment Questionnaire Disability Index (HAQ DI), and CRP level
Disease activity scale in 28 joints (DAS-28) | week 12
  Scale assessing severity of rheumatoid arthritis based on number of tender, swollen joints, erythrocyte sedimentation rate (ESR) levels, and patient self-assessment of his condition (global health assessment). Whereas "28" describes the number of different joints including in the measurement: proximal interphalangeal joints (10 joints), metacarpophalangeal joints (10), wrists (2), elbows (2), shoulders (2), knees (2).

SECONDARY OUTCOMES:
GRK2 expression | week 12
  GRK2 expression in serum
TNF-α | week 12
  Serum level Tumor necrosis factor- alpha (TNF-α)
Inteleukins | 12 weeks
  Serum levels of Interleukins (IL) IL-17, IL-1β , IL-6 & IL-10
CRP | 12 weeks
  Serum level of C-reactive protein (CRP)
Drug Adverse effects | 12 weeks
  Adverse effect incidence: adverse effect will be reported by patients or their caregivers and recorded by investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF